CLINICAL TRIAL: NCT02276274
Title: A Randomized, Open-label, Crossover Study to Determine the Effect of Food on the Pharmacokinetics of Single Oral Dose Administration of a Fixed-Dose Combination of SYR-322 and Metformin Hydrochloride in Healthy Adult Male Subjects
Brief Title: Effect of Food on the Pharmacokinetics of Single Oral Dose Administration of a Fixed-Dose Combination of SYR-322 and Metformin Hydrochloride in Healthy Adult Male Subjects
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Basic Science
Other Study IDs: SYR-322-MET/CPH-002; U1111-1157-8500 (Other: UTN); JapicCTI-142584 (Registry Identifier: JapicCTI (Japan))
Record Dates: First submitted 2014-06-26; First posted 2014-10-28 (Estimated); Results first posted 2015-06-29 (Estimated); Last update posted 2023-09-21 (Actual); Status verified 2023-08

CONDITIONS: Clinical Pharmacology

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Fasted dosing followed by fed dosing (Experimental): Oral administration
  Interventions: Drug: SYR-322-MET
- Fed dosing followed by fasted dosing (Experimental): Oral administration
  Interventions: Drug: SYR-322-MET

INTERVENTIONS:
Drug: SYR-322-MET — Oral administration of SYR-322-MET

SUMMARY:
This is a randomized, open-label, crossover study to determine the effect of food when a combination tablet of SYR-322 and metformin hydrochloride ( hereinafter referred to as SYR-322-MET tablet) is orally administered under fasting conditions in the morning or after breakfast in Japanese healthy adult male subjects.

DETAILED DESCRIPTION:
The primary objective of this clinical trial is to determine the effect of food on the pharmacokinetics of single oral dose administration of SYR-322-MET tablets in Japanese healthy adult male subjects

ELIGIBILITY:
Inclusion Criteria:

1. In the opinion of the investigator or subinvestigator, the subject is capable of understanding and complying with protocol requirements.
2. The subject signs and dates a written, informed consent form prior to the initiation of any study procedures.
3. The subject is a Japanese healthy adult male.
4. The subject is aged 20 to 35 years, inclusive, at the time of informed consent.
5. The subject has a body weight of 50 kg or more with a BMI of ≥18.5 kg/m2 and <25.0 kg/m2 at screening.

Exclusion Criteria:

1. The subject has received any investigational compound within 16 weeks (112 days) prior to the start of study drug administration in Period 1.
2. The subject has received SYR-322 or metformin hydrochloride in a previous clinical study or as a therapeutic agent.
3. The subject is an immediate family member, study site employee, or is in a dependant relationship with a study site employee who is involved in the conduct of this study (eg, spouse, parent, child, sibling) or may consent under duress.
4. The subject has uncontrolled, clinically significant neurologic, cardiovascular, pulmonary, hepatic, renal, metabolic, gastrointestinal, urologic, or endocrine disease or other abnormality, which may impact the ability of the subject to participate or potentially confound the study results.
5. The subject has a known hypersensitivity to drugs.
6. The subject has a positive urine drug result for drugs of abuse (defined as any illicit drug use) at screening.
7. The subject has a history of drug abuse or history of alcohol abuse within 2 years prior to the screening visit or unwilling to agree to abstain from alcohol and drugs throughout the study.
8. Subject has taken any excluded medication, supplements, or food products during the time periods listed in the Excluded Medications and Dietary Products table.
9. Subject has evidence of current cardiovascular, central nervous system, hepatic, hematopoietic disease, renal dysfunction, metabolic or endocrine dysfunction, serious allergy, asthma, hypoxemia, hypertension, seizures, or allergic skin rash. There is any finding in the subject's medical history, physical examination, or safety laboratory tests giving reasonable suspicion of a disease that would contraindicate taking DPP-4 inhibitors or biguanides, or a similar drug in the same class, or that might interfere with the conduct of the study. This includes, but is not limited to, peptic ulcer disease, seizure disorders, and cardiac arrhythmias.
10. The subject has current or recent [within 24 weeks (168 days) prior to the initiation of study treatment in Period 1] gastrointestinal disease that would be expected to influence the absorption of drugs (i.e., a history of malabsorption, esophageal reflux, peptic ulcer disease, erosive esophagitis, frequent [more than once per week] occurrence of heartburn, or any surgical intervention [e.g., cholecystectomy]).
11. The subject has a history of cancer.
12. The subject has a positive test result for hepatitis B surface antigen (HBsAg), hepatitis C antibody (HCV), human immunodeficiency virus (HIV) antibody/antigen, or serological reactions for syphilis at screening.
13. The subject has poor peripheral venous access.
14. The subject has undergone whole blood collection of at least 200 mL within 4 weeks (28 days) or at least 400 mL within 12 weeks (84 days) prior to the start of study medication administration Period 1.
15. The subject has undergone whole blood collection of at least 800 mL in total within 52 weeks (364 days) prior to the start of study medication administration in Period 1.
16. The subject has undergone blood component collection within 2 weeks (14 days) prior to the start of study medication administration in Period 1.
17. The subject has a screening or prior to the start of study medication administration on Day 1 in Period 1 hemoglobin level <12.5 g/dL.
18. The subject has a screening or prior to the start of study medication administration on Day 1 in Period 1 abnormal (clinically significant) 12-lead ECG.
19. Subject has abnormal screening or prior to the start of study medication administration on Day 1 in Period 1 laboratory values that suggest a clinically significant underlying disease or subject with the following lab abnormalities: ALT and/or AST >1.5 the upper limits of normal.
20. Subject who, in the opinion of the investigator, is unlikely to comply with the protocol or is unsuitable for any other reason.

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2014-06; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: General Manager, Study Director — Takeda Pharmaceutical Company Limited (Japan)
Locations (1):
- Fukuoka, Fukuoka, Japan

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 1 investigative site in Japan from 21 June 2014 to 22 July 2014.
Pre-assignment Details: Healthy participants were enrolled in 1 of 2 treatment groups: SYR-322-MET fasted followed by SYR-322-MET fed; SYR-322-MET fed followed by SYR-322-MET fasted.
Groups:
- SYR-322-MET Fasted Followed by SYR-322-MET Fed: A single dose of SYR-322 25 milligram (mg) and metformin hydrochloride 500 mg in 1 tablet, orally under fasted condition on Day 1 of first intervention period, followed by at least 15 days of washout period, followed by a single dose of SYR-322 25 mg and metformin hydrochloride 500 mg in 1 tablet, orally under fed condition on Day 1 of second intervention period.
- SYR-322-MET Fed Followed by SYR-322-MET Fasted: A single dose of SYR-322 25 mg and metformin hydrochloride 500 mg in 1 tablet, orally under fed condition on Day 1 of first intervention period, followed by at least 15 days of washout period, followed by a single dose of SYR-322 25 mg and metformin hydrochloride 500 mg in 1 tablet, orally under fasted condition on Day 1 of second intervention period.
Period: First Intervention Period
Arm/Group | SYR-322-MET Fasted Followed by SYR-322-MET Fed | SYR-322-MET Fed Followed by SYR-322-MET Fasted
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Washout Period (at Least 15 Days)
Arm/Group | SYR-322-MET Fasted Followed by SYR-322-MET Fed | SYR-322-MET Fed Followed by SYR-322-MET Fasted
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0
Period: Second Intervention Period
Arm/Group | SYR-322-MET Fasted Followed by SYR-322-MET Fed | SYR-322-MET Fed Followed by SYR-322-MET Fasted
Started | 6 | 6
Completed | 6 | 6
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Pharmacokinetic analysis set: subset of participants who received the investigational product, satisfied the minimum requirements of the protocol with no significant deviations, and were assessable for pharmacokinetics.
Groups:
- Total: Total of all reporting groups
Arm/Group | SYR-322-MET Fasted Followed by SYR-322-MET Fed | SYR-322-MET Fed Followed by SYR-322-MET Fasted | Total
Number analyzed (Participants) | 6 | 6 | 12
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (1.94) | 27.2 (6.43) | 25.2 (4.99)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 6 | 6 | 12
height [Mean (Standard Deviation); unit: centimeters (cm)] | 168.5 (6.98) | 175.7 (6.68) | 172.1 (7.51)
Weight [Mean (Standard Deviation); unit: kilogram (kg)] | 61.17 (8.373) | 65.40 (6.425) | 63.28 (7.451)
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kilogram per square meter (kg/m^2)] | 21.48 (1.878) | 21.15 (0.869) | 21.32 (1.406)
Smoking Classification [Number; unit: participants]
  Never Smoked | 2 | 1 | 3
  Current Smoker | 3 | 3 | 6
  Ex-Smoker | 1 | 2 | 3
Alcohol Classification [Number; unit: participants]
  Drank Every Day | 0 | 0 | 0
  Drank a Few Days per Week | 0 | 0 | 0
  Drank a Few Days per Month | 4 | 3 | 7
  No | 2 | 3 | 5
Caffeine Classification [Number; unit: participants]
  Took Caffeine | 2 | 1 | 3
  Did not take Caffeine | 4 | 5 | 9

OUTCOME MEASURES:

1. Primary Outcome: AUC (0-72): Area Under the Plasma Concentration-time Curve From Time 0 to 72 Hours Postdose for Unchanged SYR-322 (SYR-322Z)
Description: AUC (0-72) is measure of area under the curve from time 0 to 72 hours post dose.
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48, and 72 hours postdose
Population: Pharmacokinetic set: subset of participants who received the investigational product, satisfied the minimum requirements of the protocol with no significant deviations, and were assessable for pharmacokinetics.
Measure: Mean (Standard Deviation); unit: nanogram*milliliter per hour (ng*hr/mL)
Groups:
- SYR-322-MET Fasted: SYR-322 25 mg and metformin hydrochloride 500 mg in 1 tablet, orally, under fasted condition on Day 1 of either first or second intervention period.
- SYR-322-MET Fed: SYR-322 25 mg and metformin hydrochloride 500 mg in 1 tablet, orally, under fed condition on Day 1 of either first or second intervention period.
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
nanogram*milliliter per hour (ng*hr/mL) | 1494.9 (159.42) | 1472.8 (172.59)
Statistical Analysis 1: Comparison: SYR-322-MET Fasted vs SYR-322-MET Fed; Test type: Superiority or Other; Least Squares Mean Difference = -0.0164, 90% CI 2-sided [-0.0592 to 0.0264] — Analysis of variance (ANOVA) was performed on log-transformed values of AUC (0-72) with regimen, treatment group (treatment sequence), and treatment period as fixed effects

2. Primary Outcome: AUC (0-tlqc): Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for SYR-322Z
Description: AUC (0-tlqc) is a measure of total plasma exposure to the drug from Time 0 to Time of the Last Quantifiable Concentration (AUC [0-tlqc]).
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 1494.9 (159.42) | 1472.8 (172.59)
Statistical Analysis 1: Comparison: SYR-322-MET Fasted vs SYR-322-MET Fed; Test type: Superiority or Other; Least Squares Mean Difference = -0.0164, 90% CI 2-sided [-0.0592 to 0.0264] — ANOVA was performed on log-transformed values of AUC (0-tlqc) with regimen, treatment group (treatment sequence), and treatment period as fixed effects

3. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for SYR-322Z
Description: Maximum observed plasma concentration (Cmax) is the peak plasma concentration of a drug after administration, obtained directly from the plasma concentration-time curve.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
ng/mL | 154.9 (38.72) | 173.4 (38.45)
Statistical Analysis 1: Comparison: SYR-322-MET Fasted vs SYR-322-MET Fed; Test type: Superiority or Other; Least Squares Mean Difference = 0.1182, 90% CI 2-sided [-0.0405 to 0.2769] — ANOVA was performed on log-transformed values of Cmax with regimen, treatment group (treatment sequence), and treatment period as fixed effects

4. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for SYR-322Z
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Median (Full Range); unit: hour (hr)
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hour (hr) | 3.000 [2.00 to 4.00] | 1.00 [0.50 to 3.00]

5. Primary Outcome: AUC (0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for SYR-322Z
Description: AUC (0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 1555.0 (167.20) | 1536.8 (187.33)
Statistical Analysis 1: Comparison: SYR-322-MET Fasted vs SYR-322-MET Fed; Test type: Superiority or Other; Least Squares Mean Difference = -0.0139, 90% CI 2-sided [-0.0598 to 0.0320] — ANOVA was performed on log-transformed values of AUC (0-inf) with regimen, treatment group (treatment sequence), and treatment period as fixed effects

6. Primary Outcome: Apparent Terminal Elimination Rate Constant (λz) for SYR-322Z
Description: Terminal elimination rate constant, calculated as the negative of the slope of the log-linear regression of the natural logarithm concentration-time curve during the terminal phase.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr^-1
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr^-1 | 0.03912 (0.0046649) | 0.03673 (0.0053316)

7. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) for SYR-322Z
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr | 17.94 (2.0527) | 19.24 (2.8931)

8. Primary Outcome: Apparent Clearance After Extra Vascular Administration (CL/F) for SYR-322Z
Description: CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided AUC (0-inf), expressed in liter/hour (L/hr).
Time Frame: 3 hours prior to administration, and at 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, 48 and 72 hours after administration
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
L/hr | 16.24 (1.6898) | 16.52 (2.2647)

9. Primary Outcome: Mean Residence Time (MRT) for SYR-322Z
Description: Mean residence time (MRT) calculated as area under the first moment plasma concentration-time curve (AUMC [0-inf]) divided by AUC (0-inf). (AUMC [0-inf]) is the area under the first moment plasma concentration-time curve from time 0 to infinity.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr | 18.06 (1.4216) | 17.72 (2.1696)

10. Primary Outcome: MRT (0-tlqc): Mean Residence Time From Time 0 to Time of the Last Quantifiable Concentration (Tlqc) for SYR-322Z
Description: MRT (0-tlqc) is a measure of the mean residence time from time 0 to time of the last quantifiable concentration (tlqc) calculated as MRT (0-tlqc) =AUMC (0-tlqc)/AUC (0-tlqc). AUMC (0-tlqc) is the area under the first moment plasma concentration-time curve from time 0 to time of the last quantifiable concentration (tlqc), calculated using the linear trapezoidal rule.
Time Frame: as for outcome 1
Population: as for baseline characteristics
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr | 14.84 (1.2056) | 14.17 (1.1703)

11. Primary Outcome: AUC (0-72): Area Under the Plasma Concentration-time Curve From Time 0 to 72 Hours Post Dose for SYR-322 Metabolites M-I and M-II
Description: AUC (0-72) is measure of area under the curve from time 0 to 72 hours post dose.
Time Frame: as for outcome 1
Population: Pharmacokinetic set: subset of participants who received the investigational product, satisfied the minimum requirements of the protocol with no significant deviations, and were assessable for pharmacokinetics of each of the SYR-322 metabolites.
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL
  M-I | 9.49 (7.746) | 8.28 (6.862)
  M-II | 39.18 (26.439) | 37.00 (26.048)

12. Primary Outcome: AUC (0-tlqc): Area Under the Plasma Concentration-time Curve From Time 0 to the Time of the Last Quantifiable Concentration for SYR-322 Metabolites M-I and M-II
Description: as for outcome 2
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL
  M-I | 8.93 (7.828) | 7.72 (6.906)
  M-II | 38.48 (26.579) | 36.00 (25.861)

13. Primary Outcome: MRT (0-tlqc): Mean Residence Time From Time 0 to Time of the Last Quantifiable Concentration (Tlqc) for SYR-322 Metabolites M-I and M-II
Description: as for outcome 10
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr
  M-I (n= 11, 11) | 17.95 (6.3662) | 17.75 (6.7278)
  M-II (n=12, 12) | 10.88 (1.6364) | 10.45 (1.7285)

14. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for SYR-322 Metabolites M-I and M-II
Description: as for outcome 3
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
ng/mL
  M-I | 0.42 (0.295) [1.50 to 4.00] | 0.40 (0.319) [1.00 to 4.00]
  M-II | 4.18 (3.052) [3.00 to 4.00] | 3.58 (2.525) [1.50 to 3.00]

15. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for SYR-322 Metabolites M-I and M-II
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Median (Full Range); unit: hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr
  M-I (n = 11, 11) | 3.000 (9.168) [1.50 to 4.00] | 1.500 (6.369) [1.00 to 4.00]
  M-II (n = 12, 12) | 3.000 (27.226) [3.00 to 4.00] | 2.500 (26.671) [1.50 to 3.00]

16. Primary Outcome: AUC (0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for SYR-322 Metabolites M-I and M-II
Description: AUC (0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL
  M-I (n = 9, 9) | 15.86 (9.168) | 14.53 (6.369)
  M-II (n = 12, 12) | 40.28 (27.226) | 38.01 (26.671)

17. Primary Outcome: Apparent Terminal Elimination Rate Constant (λz) for SYR-322 Metabolites M-I and M-II
Description: as for outcome 6
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hr^-1
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr^-1
  M-I (n = 9, 9) | 0.02711 (0.0039065) | 0.02708 (0.0081278)
  M-II (n = 12, 12) | 0.06458 (0.023460) | 0.06651 (0.021985)

18. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) for SYR-322 Metabolites M-I and M-II
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr
  M-I (n = 9, 9) | 26.09 (3.9939) | 31.39 (22.996)
  M-II (n = 12, 12) | 12.43 (5.4904) | 11.70 (4.5855)

19. Primary Outcome: Mean Residence Time (MRT) for SYR-322 Metabolites M-I and M-II
Description: Mean residence time (MRT) calculated as area under the first moment plasma concentration-time curve (AUMC [0-inf]) divided by AUC (0-inf). AUMC (0-inf) is the area under the first moment plasma concentration-time curve from time 0 to infinity.
Time Frame: as for outcome 1
Population: as for outcome 11
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr
  M-I (n = 9, 9) | 39.87 (6.1272) | 49.97 (38.556)
  M-II (n = 12, 12) | 13.93 (2.2797) | 13.81 (2.1894)

20. Primary Outcome: AUC (0-48): Area Under the Plasma Concentration-time Curve From Time 0 to 48 Hours Postdose for Metformin
Description: AUC (0-48) is measure of area under the curve from time 0 to 48 hours post dose.
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 9157.3 (1684.53) | 8991.8 (1284.97)
Statistical Analysis 1: Comparison: SYR-322-MET Fasted vs SYR-322-MET Fed; Test type: Superiority or Other; Least Squares Mean Difference = -0.0140, 90% CI 2-sided [-0.0918 to 0.0638] — ANOVA was performed on log-transformed values of AUC (0-48) with regimen, treatment group (treatment sequence), and treatment period as fixed effects

21. Primary Outcome: AUC (0-tlqc): Area Under the Plasma Concentration-Time Curve From Time 0 to the Time of the Last Quantifiable Concentration for Metformin
Description: as for outcome 2
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 9038.8 (1661.09) | 8853.8 (1271.92)
Statistical Analysis 1: Comparison: SYR-322-MET Fasted vs SYR-322-MET Fed; Test type: Superiority or Other; Least Squares Mean Difference = -0.0164, 90% CI 2-sided [-0.0934 to 0.0605] — [estimate comment as in outcome 2, analysis 1]

22. Primary Outcome: MRT (0-tlqc): Mean Residence Time From Time 0 to Time of the Last Quantifiable Concentration (Tlqc) for Metformin
Description: as for outcome 10
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr | 5.697 (0.75798) | 5.697 (0.58215)

23. Primary Outcome: Cmax: Maximum Observed Plasma Concentration for Metformin
Description: as for outcome 3
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng/mL
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
ng/mL | 1473.3 (300.19) | 1251.7 (164.03)
Statistical Analysis 1: Comparison: SYR-322-MET Fasted vs SYR-322-MET Fed; Test type: Superiority or Other; Least Squares Mean Difference = -0.1518, 90% CI 2-sided [-0.2356 to -0.0680] — [estimate comment as in outcome 3, analysis 1]

24. Primary Outcome: Tmax: Time to Reach the Maximum Plasma Concentration (Cmax) for Metformin
Description: Tmax: Time to reach the maximum plasma concentration (Cmax), equal to time (hours) to Cmax.
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: as for outcome 1
Measure: Median (Full Range); unit: hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr | 3.000 [0.50 to 4.00] | 3.000 [0.50 to 4.00]

25. Primary Outcome: AUC (0-inf): Area Under the Plasma Concentration-time Curve From Time 0 to Infinity for Metformin
Description: AUC (0-inf) is a measure of total plasma exposure to the drug from time zero extrapolated to infinity.
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ng*hr/mL
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
ng*hr/mL | 9195.3 (1669.37) | 8997.4 (1289.67)
Statistical Analysis 1: Comparison: SYR-322-MET Fasted vs SYR-322-MET Fed; Test type: Superiority or Other; Least Squares Mean Difference = -0.0179, 90% CI 2-sided [-0.0950 to 0.0591] — [estimate comment as in outcome 5, analysis 1]

26. Primary Outcome: Apparent Terminal Elimination Rate Constant (λz) for Metformin
Description: as for outcome 6
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr^-1
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr^-1 | 0.1366 (0.028295) | 0.1638 (0.027820)

27. Primary Outcome: Terminal Phase Elimination Half-life (T1/2) for Metformin
Description: Terminal phase elimination half-life (T1/2) is the time required for half of the drug to be eliminated from the plasma.
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr | 5.290 (1.1735) | 4.338 (0.70681)

28. Primary Outcome: Apparent Clearance After Extra Vascular Administration (CL/F) for Metformin
Description: CL/F is apparent clearance of the drug from the plasma, calculated as the drug dose divided AUC (0-inf), expressed in L/hr.
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
L/hr | 55.84 (9.0078) | 56.75 (9.1099)

29. Primary Outcome: Mean Residence Time (MRT) for Metformin
Description: as for outcome 19
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hr | 6.213 (0.88315) | 6.097 (0.63435)

30. Primary Outcome: Urinary Excretion Ratio of SYR-322Z From 0 to 12 Hours Postdose
Description: Cumulative urinary excretion ratio of unchanged SYR-322 was calculated as the percentage of SYR-322 dose.
Time Frame: 0 to 12 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of dose | 42.609 (4.9985) | 45.028 (6.9388)

31. Primary Outcome: Urinary Excretion Ratio of SYR-322Z From 0 to 24 Hours Postdose
Description: Cumulative urinary excretion ratio of unchanged SYR-322 was calculated as the percentage of SYR-322 dose.
Time Frame: 0 to 24 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of dose | 58.618 (4.0606) | 59.886 (6.5474)

32. Primary Outcome: Urinary Excretion Ratio of SYR-322Z From 0 to 48 Hours Postdose
Description: Cumulative urinary excretion ratio of unchanged SYR-322 was calculated as the percentage of SYR-322 dose.
Time Frame: 0 to 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of dose | 70.200 (3.8051) | 71.148 (6.4985)

33. Primary Outcome: Urinary Excretion Ratio of SYR-322Z From 0 to 72 Hours Postdose
Description: Cumulative urinary excretion ratio of unchanged SYR-322 was calculated as the percentage of SYR-322 dose.
Time Frame: 0 to 72 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of dose | 73.728 (3.9140) | 74.547 (6.4048)

34. Primary Outcome: Urinary Excretion Ratio of SYR-322 Metabolites M-I and M-II From 0 to 12 Hours Postdose
Description: Cumulative urinary excretion ratio of SYR-322 metabolites M-I and M-II was calculated as the percentage of SYR-322 dose.
Time Frame: 0 to 12 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of dose
  M-I | 0.235 (0.1393) | 0.234 (0.1719)
  M-II | 1.202 (0.8060) | 1.145 (0.7826)

35. Primary Outcome: Urinary Excretion Ratio of SYR-322 Metabolites M-I and M-II From 0 to 24 Hours Postdose
Description: Cumulative urinary excretion ratio of SYR-322 metabolites M-I and M-II was calculated as the percentage of SYR-322 dose.
Time Frame: 0 to 24 hours post dose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of dose
  M-I | 0.394 (0.2386) | 0.363 (0.2482)
  M-II | 1.562 (1.0106) | 1.502 (0.9879)

36. Primary Outcome: Urinary Excretion Ratio of SYR-322 Metabolites M-I and M-II From 0 to 48 Hours Postdose
Description: Cumulative urinary excretion ratio of SYR-322 metabolites M-I and M-II was calculated as the percentage of SYR-322 dose.
Time Frame: 0 to 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of dose
  M-I | 0.535 (0.3441) | 0.495 (0.3352)
  M-II | 1.788 (1.1384) | 1.732 (1.1284)

37. Primary Outcome: Urinary Excretion Ratio of SYR-322 Metabolites M-I and M-II From 0 to 72 Hours Postdose
Description: Cumulative urinary excretion ratio of SYR-322 metabolites M-I and M-II was calculated as the percentage of SYR-322 dose.
Time Frame: 0 to 72 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of dose
  M-I | 0.588 (0.3884) | 0.536 (0.3816)
  M-II | 1.853 (1.1929) | 1.796 (1.1696)

38. Primary Outcome: Urinary Excretion Ratio of Metformin From Time 0 to 12 Hours Postdose
Description: Cumulative urinary excretion ratio of metformin was calculated as the percentage of metformin dose.
Time Frame: 0 to 12 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of dose | 45.143 (7.7692) | 44.809 (7.4874)

39. Primary Outcome: Urinary Excretion Ratio of Metformin From 0 to 24 Hours Postdose
Description: Cumulative urinary excretion ratio of metformin was calculated as the percentage of metformin dose.
Time Frame: 0 to 24 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of dose | 50.078 (7.5995) | 49.923 (7.5189)

40. Primary Outcome: Urinary Excretion Ratio of Metformin From 0 to 48 Hours Postdose
Description: Cumulative urinary excretion ratio of metformin was calculated as the percentage of metformin dose.
Time Frame: 0 to 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: percentage of dose
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of dose | 50.626 (7.6377) | 50.067 (7.6636)

41. Primary Outcome: CLr: Renal Clearance of SYR-322Z
Description: CLr is a measure of apparent clearance of the drug from the urine. The clearance is the rate at which waste substances are cleared from the blood.
Time Frame: as for outcome 1
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
L/hr | 11.96 (1.2071) | 12.33 (2.2296)

42. Primary Outcome: CLr: Renal Clearance of Metformin
Description: CLr is a measure of apparent clearance of the drug from the urine.
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8, 12, 16, 24, 36, and 48 hours postdose
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: L/hr
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
L/hr | 27.88 (4.1525) | 28.34 (6.3364)

43. Secondary Outcome: Inhibition Rate of Dipeptidyl-peptidase-4 (DPP-4) Activity
Description: DPP-4 activity and inhibition rate of DPP-4 activity was assessed from the plasma samples collected from the participants. Inhibition of DPP-4 enzyme was used to determine the antihyperglycemic activity of the investigational product.
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours postdose
Population: Pharmacodynamic analysis set: subset of participants who received the investigational product, satisfied the minimum requirements of the protocol with no significant deviations, and were assessable for pharmacodynamics.
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of inhibition
  Predose | 0.00 (0.000) | 0.00 (0.000)
  0.25 hour | 68.00 (26.599) | 57.99 (32.209)
  0.5 hour | 85.65 (17.721) | 90.31 (7.533)
  1 hour | 91.05 (4.070) | 95.27 (2.371)
  1.5 hour | 91.85 (2.342) | 95.79 (0.710)
  2 hour | 93.63 (2.028) | 95.58 (0.542)
  3 hour | 95.52 (1.528) | 94.71 (0.611)
  4 hour | 94.88 (1.216) | 93.78 (0.877)
  6 hour | 93.04 (0.708) | 92.06 (0.880)
  8 hour | 91.78 (0.890) | 90.51 (1.071)
  24 hour | 81.74 (2.235) | 81.38 (2.614)

44. Secondary Outcome: DPP-4 Activity
Description: DPP-4 activity was assessed from the plasma samples collected from the participants.
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours postdose
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: nanomole/minute/milliliter (nmoL/min/mL)
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
nanomole/minute/milliliter (nmoL/min/mL)
  Predose | 7.8167 (0.85551) | 7.8492 (0.99173)
  0.25 hour | 2.5833 (2.37291) | 3.4518 (2.86390)
  0.5 hour | 1.1944 (1.64100) | 0.7823 (0.66267)
  1 Hour | 0.7122 (0.39573) | 0.3737 (0.21081)
  1.5 Hour | 0.6366 (0.19955) | 0.3312 (0.07085)
  2 hours | 0.5003 (0.17621) | 0.3475 (0.05993)
  3 hours | 0.3575 (0.14924) | 0.4128 (0.06132)
  4 hours | 0.3977 (0.09285) | 0.4873 (0.08441)
  6 hours | 0.5423 (0.07347) | 0.6196 (0.08548)
  8 hours | 0.6422 (0.09457) | 0.7425 (0.11652)
  24 hours | 1.4275 (0.22071) | 1.4550 (0.24055)

45. Secondary Outcome: AUC (0-24): Area Under the Inhibition Rate of Plasma DPP-4 Activity-time Curve From Time 0 to 24 Hours
Description: Area under the inhibition rate of plasma DPP-4 activity-time curve from time 0 to 24 hours was determined from the inhibition-time curve.
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours postdose
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: percentage of inhibition*hour
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of inhibition*hour | 2114.62 (30.355) | 2100.74 (27.297)

46. Secondary Outcome: Emax: Maximum Inhibition Rate of Plasma DPP-4 Activity
Description: Maximum inhibition rate of plasma DPP-4 activity was determined from the inhibition-time curve.
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours postdose
Population: as for outcome 43
Measure: Mean (Standard Deviation); unit: percentage of inhibition
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
percentage of inhibition | 96.10 (1.022) | 96.33 (0.779)

47. Secondary Outcome: Tmax: Time to Reach Emax
Description: Time to reach Emax for the first time was determined from the inhibition-time curve.
Time Frame: 3 hours prior to administration (predose) and 0.25, 0.5, 1, 1.5, 2, 3, 4, 6, 8 and 24 hours postdose
Population: as for outcome 43
Measure: Median (Full Range); unit: hour
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
hour | 3.000 [2.00 to 4.00] | 1.000 [0.50 to 2.00]

48. Secondary Outcome: Number of Participants Reporting 1 or More Treatment-emergent Adverse Events
Description: An Adverse Event (AE) is defined as any untoward medical occurrence in a clinical investigation participant administered a drug; it does not necessarily have to have a causal relationship with this treatment. An AE can therefore be any unfavorable and unintended sign (eg, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A treatment-emergent adverse event (TEAE) is defined as an adverse event with an onset that occurs after receiving study drug.
Time Frame: Baseline up to the day of discharge (Day 4) in the second intervention period
Population: Safety analysis set: All participants who receive at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

49. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Vital Signs
Description: Vital signs included body temperature (infra-axillary), supine blood pressure resting more than 5 minutes (systolic and diastolic [Millimeters of mercury]), respiratory rate and pulse (beats per minute). Clinically significant change in vital signs observed at any time point are reported.
Time Frame: 3 hours prior to administration (predose) and 2, 24 and 72 hours postdose
Population: Safety analysis set: All participants who receive at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

50. Secondary Outcome: Number of Participants With Clinically Significant Change From Baseline in Body Weight
Description: Clinically significant change participant's body weight observed at any time point are reported.
Time Frame: 3 hours prior to administration (predose), 24 and 72 hours postdose
Population: Safety analysis set: All participants who receive at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

51. Secondary Outcome: Number of Participants With Significant Change From Baseline in Electrocardiograms
Description: Clinically significant change in electrocardiograms observed at any time point are reported.
Time Frame: 3 hours prior to administration (predose) and 2, 24 and 72 hours postdose
Population: Safety analysis set: All participants who receive at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

52. Secondary Outcome: Number of Participants With Laboratory-related Treatment Emergent Adverse Events (TEAEs)
Description: Laboratory assessments included hematology, serum chemistry and urinalysis. Any laboratory-related TEAE reported at any time point were reported in this measure.
Time Frame: 3 hours prior to administration (predose), 24 and 72 hours postdose
Population: Safety analysis set: All participants who receive at least one dose of study medication.
Measure: Number; unit: participants
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Number analyzed (Participants) | 12 | 12
participants | 0 | 0

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events are adverse events that started after the first dose of the study drug and up to the day of discharge (Day 4) in the second intervention period.
Description: At each visit the investigator had to document any occurrence of adverse events and abnormal laboratory findings. Any event spontaneously reported by the participant or observed by the investigator was recorded, irrespective of the relation to study treatment.
Arm/Group | SYR-322-MET Fasted | SYR-322-MET Fed
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/12
Other Adverse Events (participants affected / at risk) | 0/12 | 0/12

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The first study related publication will be a multi-center publication submitted within 24 months after conclusion or termination of a study at all sites. After such multi site publication, all proposed site publications and presentations will be submitted to sponsor for review 60 days in advance of publication. Site will remove Sponsor confidential information unrelated to study results. Sponsor can delay a proposed publication for another 60 days to preserve intellectual property.